CLINICAL TRIAL: NCT04422847
Title: Use of Computer Aided Design and 3D Printing for Anesthesiology Management in a Pediatric Patient With Cleft Facial Defect
Acronym: 3D obturator
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Collaborators: Brno University of Technology (Other); Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3D Obturator
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cleft Lip and Palate
Keywords: 3D print; Cleft surgery; Paediatric; Airway
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Intervention Model Description: Patient will be randomized according to the interventional and control goup according to the day of surgery. The allocation between the groups will be 1:1
Masking Description: No masking will be included
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (3D protective obturator) (Experimental): Patients enrolled in the intervention group will have an intraoral scan of the palate, alveolar arch, and upper vestibular area before surgery. Based on this 3D visualization of precise anatomical conditions in the oral cavity, a form (negative unique impression of the upper jaw and palato-alveolar conditions) for casting of a protective obturator (splint), used during intubation to cover the defect of the alveolar arch and palate will be created on a 3D printer, in cooperation with the Faculty of Mechanical Engineering (Department of Mechanics of Bodies, Mechatronics and Biomechanics) of Brno University of Technology. For the production of the obturator, a silicone certified for use in the oral cavity will be used.
  Interventions: Device: 3D obturator
- control group (No Intervention): The standard procedure without the 3D obturator.

INTERVENTIONS:
Device: 3D obturator — Based on this 3D visualization of precise anatomical conditions in the oral cavity, a form (negative unique impression of the upper jaw and palato-alveolar conditions) for casting of a protective obturator (splint), used during intubation to cover the defect of the alveolar arch and palate will be created on a 3D printer
  Other Names: 3D printer obturator
  Arms: intervention group (3D protective obturator)

SUMMARY:
Congenital malformations of the orofacial area are the most common congenital malformations in children with an incidence of 1.8 children with orofacial cleft per 1000 healthy births in the Czech Republic. The care of children with cleft facial defects is multidisciplinary, centralized and takes place from birth to adulthood. At the University Hospital Brno, the treatment for patients with orofacial cleft is provided by the Cleft Center (CC) of the University Hospital Brno. The main specialties that form the basis of CC include plastic surgery, pediatric anesthesiology and neonatology. Patients with facial cleft defects are divided into 2 main groups based on the embryological causes of clefts: 1/ patients with cleft lip, jaw with or without cleft palate (total cleft) and 2/ patients with isolated cleft soft and hard palate. Anesthesia in children with orofacial clefts is specific not only to the age of the patients, but mainly to the cleft itself. Anesthesiology management, and especially intubation of these patients, are often difficult due to the nature of the defect with high incidence of complications such as difficult airway, desaturation, laryngospasm or bradycardia. In addition, tissue damage including soft tissue of the lip, alveolar arch, palate and nasal septum as well as skeleton of the premaxilla and nasal septum during intubation is seen in approximately 90% of patients. To facilitate intubation, improve anesthesiology management and safety of pediatric patients with orofacial cleft, we will develop an individualized protective tray from a silicone material, that will be used during intubation to cover the defect of the alveolar arch and palate. A mold for casting of a protective tray, will be created on a 3D printer on bases of 3D scan. Use of the protective tray would facilitate intubation, decrease anesthesiologic complications and protect soft and hard tissues of the cleft palate and upper jaw during intubation.

DETAILED DESCRIPTION:
After approval by the Ethics Committee of the Brno University Hospital and registration at clinicaltrials.gov, the study will include patients meeting inclusive criteria for whom primary surgery for a cleft facial defect will be indicated.

Patients will be divided into two groups based on the type of surgery. Group 1 will include patients with unilateral or bilateral cleft lip and alveolus (U/BCLA) or unilateral or bilateral cleft lip, alveolus and palate (total cleft; U/BCLAP) who underwent primary lip reconstruction within 0-3 months of age. Group 2 will include patients with isolated cleft palate (ICP) and patients with U/BCLAP who underwent primary cleft reconstruction between 6 and 18 months of age.

Patients in the pediatric plastic surgery clinic of the Department of Pediatric Surgery, Orthopedics and Traumatology will be randomized with a 1:1 allocation based on the day of operation to the intervention group (3D protective obturator) and the control group (standard procedure without the 3D obturator). Patients enrolled in the intervention group will have an intraoral scan of the palate, alveolar arch, and upper vestibular area before surgery. Based on this 3D visualization of precise anatomical conditions in the oral cavity, a form (negative unique impression of the upper jaw and palato-alveolar conditions) for casting of a protective obturator (splint), used during intubation to cover the defect of the alveolar arch and palate will be created on a 3D printer, in cooperation with the Faculty of Mechanical Engineering (Department of Mechanics of Bodies, Mechatronics and Biomechanics) of Brno University of Technology. For the production of the obturator, a silicone certified for use in the oral cavity will be used.

The main objective of the research will be to find out how the use of a protective obturator (splint) will improve the protection of tissues at the cleft site and whether intubation will be facilitated in pediatric patients with orofacial clefts with congenital atypical anatomical conditions in the oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with unilateral or bilateral cleft lip and alveolus (U/BCLA) or unilateral or bilateral cleft lip, alveolus and palate (total cleft; U/BCLAP) who underwent primary lip reconstruction within 0-3 months of age (most often at our workplace in the neonatal period)
* Pediatric patients with isolated cleft palate (ICP) and patients with unilateral or bilateral cleft lip, alveolus and palate (U/BCLAP) who underwent primary cleft reconstruction between 6 and 18 months of age.

Exclusion Criteria:

* unilateral or bilateral cleft lip without cleft alveolus
* patients with genetically confirmed syndrome disability
* orofacial cleft patients with associated congenital malformations that may affect the course of anesthesia (atresia of the choanae)
* patients with atypical clefts of the face
* patients with CLA, CLAP, ICP who underwent primary cleft lip reconstruction later than at 3 months of age
* patients with CLAP and ICP who underwent primary cleft reconstruction later than at 18 months of age
* patients with submucous cleft palate
* patients with airways secured preoperatively
* patients on artificial lung ventilation
* patients with coagulopathy, thrombocytopenia/thrombocytopathy
* patients at risk of malignant hyperthermia
* patients for whom the consent of legal representatives to the research project has not been obtained

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of oral tissue injury during intubation | Intraoperatively (after successful intubation)
  specifically presence of petechiae, bleeding or soft tissue swelling after intubation in the entire cleft defect area, possibly premaxilla fracture in total cleft patients as a result of manipulation of the laryngoscope in the oral cavity

SECONDARY OUTCOMES:
Cormack-Lehane score | Intraoperatively (during intubation)
  evaluation of the laryngoscopic image during intubation evaluated by the Cormack-Lehane score with or without the use of the protective tray. Cormack-Lehane scale range from 1 (ideal view - vocal cords) to 4 (the worst view of aditus laryngis, only the soft palate visible). For proper archiving of the intubation process, a photodocumentation of the laryngoscopic image during intubation will be taken for each patient using a video laryngoscope.

OTHER OUTCOMES:
Number of intubations attempts | Intraoperatively
  The number of intubation attempts to secure the airways (first successful intubation = first wave of end-tidal CO2) with and without the use of the protective tray will be evaluated
Incidence of associated complications | Intraoperatively
  The incidence of associated complications during induction of anesthesia - laryngospasm, bradycardia, severe desaturation < 80 % oxygen saturation oxygen saturation by pulse oximetry pulse oximetry - SpO2 will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, prof. MD., Ph.D., Study Chair — Faculty of medicince Masaryk University and University Hospital Brno
Locations (1):
- University hospital Brno, Brno, Jihomoravská Kraj, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Richtrova M, Koskova O, Marcian P, Borak L, Bonischova T, Fabian D, Janku M, Joukal M, Vymazalova K, Stourac P. Customized protective palatal obturator for intubation in newborns in cleft lip surgery: a randomized controlled trial. Ann Med. 2025 Dec;57(1):2561802. doi: 10.1080/07853890.2025.2561802. Epub 2025 Sep 22. PMID 40981509